CLINICAL TRIAL: NCT04784988
Title: Intensive Replacement Treatment in Haemophilia Patients With Synovitis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Federico II University (Other)
Responsible Party: Principal Investigator, Matteo Di Minno, Prof, Federico II University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: IISR-2020-103302
Record Dates: First submitted 2021-02-09; First posted 2021-03-05 (Actual); Last update posted 2024-03-27 (Actual); Status verified 2024-03

CONDITIONS: Hemophilia A
Keywords: Haemophilia; synovitis; ultrasound
MeSH Terms: conditions — Hemophilia A; Synovitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- PROPEL-like arm (Experimental): EHL-FVIII prophylaxis targeting a 12% FVIII through level based on PK assessment with WAPPS-Hemo
  Interventions: Drug: EHL-FVIII
- Control arm (Active Comparator): standard treatment with FVIII concentrate according to current guidelines
  Interventions: Drug: FVIII concentrate

INTERVENTIONS:
Drug: EHL-FVIII — prophylaxis with EHL-FVIII targeting a 12% FVIII through level based on PK assessment with WAPPS-Hemo
  Arms: PROPEL-like arm
Drug: FVIII concentrate — standard prophylaxis with FVIII concentrate according to current guidelines
  Arms: Control arm

SUMMARY:
Background: Joint haemorrhage represents the most common type of bleeding episode in persons with hemophilia (PwH). In the absence of an adequate prophylaxis with Factor VIII (for hemophilia A) or FIX (for hemophilia B) concentrates up to 85% of patients with severe hemophilia develop a clinically overt joint disease. Screening of early signs of arthropathy is needed. Synovitis is widely considered as one of the parameters to be taken into account for the diagnosis and the surveillance of joint impairment in PwH.

Aim: To assess if an intensive factor VIII replacement treatment is able at reverting synovitis in PwH.

Methods: The present study is a randomized, open-label, cross-over study. Among patients referred to enrolling Haemophilia Centres, consecutive patients with severe (FVIII < 1%) or severe-moderate (FVIII < 2%) haemophilia A without inhibitors will be enrolled. The present study will be organized in 2 phases.

* Phase 1 (US screening): All patients will undergo an ultrasound examination of elbows, ankles and knees to define joint status and to identify presence/absence of synovitis according to the HEAD-US system.
* Phase 2 (Intervention): Patients with US evidence of synovitis will be randomly assigned at undergoing a PK assessment with my-PK-fit to start a prophylaxis with Adynovi® targeting a 12% FVIII through level (PROPEL-like arm) or to continue ongoing standard treatment (control arm). US examination of the six joints will be repeated monthly for six months and in case of onset of symptoms that might suggest an acute bleeding episode. After six months the two treatment arm will be switched in the frame of a cross-over approach and all PwH will be followed for other 6 months The primary outcome will be represented by changes in synovial status during the intensive factor VIII replacement treatment vs standard treatment.

DETAILED DESCRIPTION:
Joint haemorrhage represents the most common type of bleeding episode in persons with hemophilia (PwH) and recurrent hemarthrosis triggers chronic arthropathy, which is the most frequent chronic complication in hemophilia patients. In the absence of an adequate prophylaxis (age at start, regimen, duration, adherence) with Factor VIII (for hemophilia A) or FIX (for hemophilia B) concentrates, up to 85% of patients with severe hemophilia develop a clinically overt joint disease.

On the other hand, some recent data suggest that, despite adequate prophylaxis a not negligible percentage of PwH develop arthropathy.

Thus, an adequate screening of early signs of arthropathy is needed. On this hand, synovitis is widely considered as one of the parameters to be taken into account for the diagnosis and the surveillance of joint impairment in PwH. Synovitis represents a key feature, potentially related to under-treatment due to insufficient therapy regimens or to a limited compliance to treatment, to pharmacokinetics variability or to demanding daily/sport activities. Accordingly, there is a general agreement on the indication to consider the presence of synovitis as a marker of disease activity in PwH.

MATERIALS AND METHODS:

Among patients referred to enrolling Haemophilia Centres (to be defined), consecutive patients with severe (FVIII < 1%) or severe-moderate (FVIII < 2%) haemophilia A without inhibitors will be enrolled according to the above reported inclusion and exclusion criteria. For each subject, a trained staff will record demographic data including age, race, ethnicity, body mass index (BMI, kg/m2). Information from medical records will also include the number of bleeding episodes and the amount of factor concentrate used during the previous 12 months for regular prophylaxis and for breakthrough bleeding episodes treatment. The present study will be organized in 2 phases.

Phase 1 (US screening): All patients will undergo an ultrasound examination of elbows, ankles and knees to define joint status and to define presence/absence of synovitis according to the HEAD-US system. Synovitis screening protocol will include examination of the olecranon recess (elbow), suprapatellar recess (knee) and anterior recess of the tibiotalar joint (ankle). For a detailed scanning protocol see Figure 1. Synovitis will be scored as absent/minimal (score 0); mild/moderate (score 1) and severe (score 2).

Phase 2 (Intervention): Patients with US evidence of synovitis will be randomly assigned at undergoing a PK assessment with WAPPS-Hemo to start a prophylaxis with any EHL-FVIII targeting a 12% FVIII through level (PROPEL-like arm) or to continue ongoing standard treatment (control arm). US examination of the six joints will be repeated monthly for six months and in case of onset of symptoms that might suggest an acute bleeding episode. For both treatment arms changes in synovitis status, the number of bleeding episodes, number of infusions and FVIII consumption will be recorded. In case of confirmed hemarthrosis an intensive treatment will be started with the ongoing treatment according to current guidelines . During the intensive treatment period, the US assessment of the affected joint will be repeated every 7 days. The intensive replacement treatment will be stopped when US will demonstrate complete resolution of intra-articular bleeding. The time to pain disappearance, the time to US evidence of bleeding resolution and the number and doses infused will be recorded for each treatment arm. Any change in prophylaxis schedule will be recorded in both treatment arms during the overall study period, and will not represent an exclusion criterion from the study.

ELIGIBILITY:
Inclusion Criteria:

1. Male patients with > 12 years of age, with severe (FVIII < 1%) or severe-moderate (FVIII < 2%) haemophilia A without inhibitors, receiving a prophylactic treatment with FVIII.
2. Evidence at ultrasound evaluation of synovitis (grade 1-2 according to HEAD-US score)
3. Signed and dated informed consent form for data collection prior to enrolment.

Exclusion Criteria:

1. Patients with bleeding disorders other than haemophilia A
2. Patients with anti-FVIII inhibitor (any titer).
3. Patients receiving on-demand treatment with FVIII
4. Patients with liver cirrhosis
5. Any condition that compromises the patient's ability to perform study-related activities or that poses a clinical contraindication to study participation.
6. Patients unwilling or unable to follow the terms of the protocol.

Ages: 12 Years to 70 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2022-03-01 (Actual); Primary Completion 2023-03-01 (Actual); Study Completion 2024-03-01 (Actual)

PRIMARY OUTCOMES:
changes in synovitis | from baseline up to 6 months
  The primary outcome of the present study is to assess if an intensive factor VIII replacement treatment is able at reverting synovitis in persons with haemophilia (PwH).

CONTACTS AND LOCATIONS:
Locations (1):
- Matteo Di Minno, Napoli, Italy